CLINICAL TRIAL: NCT05367219
Title: Composition, Hazard and Protection of Smoke From Endoscopic Gastrointestinal Surgery
Brief Title: Smoke of Endoscopic Gastrointestinal Surgery
Acronym: SEGS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: XJTU1AF2022LSK-204
Record Dates: First submitted 2022-04-24; First posted 2022-05-10 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-03

CONDITIONS: Smoke; Endoscopic Surgery; Particulate Matter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Air sterilizer (Experimental): The invesitigators will monitore smoke and try to remove the smoke with an air sterilizer during the endoscopic gastrointestinal surgery in the experimental group.
  Interventions: Device: Air sterilizer
- Control (No Intervention): The control group was monitored for smoke during the endoscopic gastrointestinal surgery without any intervention.

INTERVENTIONS:
Device: Air sterilizer — The invesitigators will try to remove the smoke with an air sterilizer during the endoscopic gastrointestinal surgery in the Air sterilizer group.
  Arms: Air sterilizer

SUMMARY:
The purpose of this project is to study the composition, hazard, and protection of smoke from endoscopic gastrointestinal surgery. The study is a single-center, prospective, randomized, controlled, cohort study. The investigators plan to enroll 80 patients who undergo endoscopic gastrointestinal surgery and 10 medical staff participating in surgery in the gastrointestinal endoscopy room of the First Affiliated Hospital of Xi'an Jiao Tong University. The investigators will randomize the included study subjects. The investigators will monitore smoke and try to remove the smoke with an air sterilizer in the Air sterilizer group. The control group was monitored for smoke without any intervention. The primary endpoint is concentration of PM2.5 in smoke from endoscopic gastrointestinal surgery, the risk factors, and the effect of air sterilizer on its removal. The secondary endpoint is the concentration of PM1.0, PM10, formaldehyde, Total Volatile Organic Compounds, CO, and CO2 in smoke from endoscopic gastrointestinal surgery, the risk factors, and the effect of air sterilizer on its removal. Other exploratory objectives include the hazards of smoke to staff in the gastrointestinal endoscopy room, and the viral content of smoke.

DETAILED DESCRIPTION:
The investigators will enroll 80 patients undergo endoscopic gastrointestinal surgery and 10 medical staff participate in surgery in the gastrointestinal endoscopy room. The patients will be randomized into the control group and the Air sterilizer group. The investigators will use air quality testing equipment to monitor the concentrations of the PM2.5, PM1.0, PM10, formaldehyde, Total Volatile Organic Compounds, CO, and CO2 of the smoke near the mouth and nose of the surgeon, cooperating nurse, and anesthesiologist, and try to remove the smoke with an air sterilizer in the Air sterilizer group. The control group was monitored for concentrations of the above ingredients in smoke without any intervention. The primary endpoint is concentration of PM2.5 in smoke during endoscopic gastrointestinal surgery, the risk factors related to surgery, and the effect of air sterilizer on its removal. The secondary endpoint is the concentration of PM1.0, PM10, formaldehyde, Total Volatile Organic Compounds, CO, and CO2 in smoke during endoscopic gastrointestinal surgery, the risk factors related to surgery, and the effect of air sterilizer on their removal. Other exploratory objectives include the hazards of smoke to staff in the gastrointestinal endoscopy room, and the viral quantitative of smoke.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo endoscopic gastrointestinal surgery and medical staff who participate in the surgery in the gastrointestinal endoscopy operating room of the First Affiliated Hospital of Xi'an Jiao Tong University
* Voluntary participation in this study

Exclusion Criteria:

* Severe liver disease
* Severe Kidney disease
* Severe cardiovascular disease
* Severe cerebrovascular disease
* Severe neuropsychiatric disease
* Unable to cooperate with the research

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-08-05 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
PM2.5 in smoke from endoscopic gastrointestinal surgery | During the surgery.
  Concentration of PM2.5 in smoke from endoscopic gastrointestinal surgery will be used by air quality testing equipment. The investigators will analyze the risk factors of PM2.5 related to surgery. The effect of air sterilizer on PM 2.5 removal will also be explored.

SECONDARY OUTCOMES:
Some other harmful substances in smoke from endoscopic gastrointestinal surgery. | During the surgery.
  Concentration of some other harmful substances in smoke from endoscopic gastrointestinal surgery including PM1.0, PM10, formaldehyde, Total Volatile Organic Compounds, CO, and CO2 in smoke will be used by air quality testing equipment. The investigators will analyze the risk factors of PM1.0, PM10, formaldehyde, Total Volatile Organic Compounds, CO, and CO2 related to surgery. The effect of air sterilizer on PM1.0, PM10, formaldehyde, Total Volatile Organic Compounds, CO, and CO2 removal will also be explored.

OTHER OUTCOMES:
Hazards of smoke to staff in the gastrointestinal endoscopy room | During the surgery and 24 hours after the surgery.
  Proportion of the endoscopy staff with smoke related adverse reactions
Viral quantitative of smoke from endoscopic gastrointestinal surgery | 40 minutes after surgery.
  In the case of patients with HBV or HIV infection, the excised tissue will be electrocuted in vitro to measure the viral quantitative in the smoke.

CONTACTS AND LOCATIONS:
Overall Officials: Shuixiang He, Study Director — First Affiliated Hospital of Xian Jiaotong University

IPD SHARING:
Plan to Share IPD: No
The invesitigators will conduct further research on endoscopic surgical smoke